CLINICAL TRIAL: NCT00949065
Title: Prospective, Double-blind, Randomised, Placebo-controlled, Cross-over Study to Investigate the Effect of Intravenous Immunoglobulins on Complex Regional Pain Syndrome (CRPS, M. Sudeck)
Brief Title: Intravenous Immunoglobulins in Complex-regional Pain Syndrome
Acronym: PAINLESS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No more interest to follow this study
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Dr. Marlene Tschernatsch, Dr., University of Giessen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-007794-23
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Complex Regional Pain Syndrome Type 1
Keywords: complex regional pain syndrome; sympathetic reflex dystrophy; intravenous immunoglobulins; autoimmune disease
MeSH Terms: conditions — Complex Regional Pain Syndromes; Reflex Sympathetic Dystrophy; Autoimmune Diseases | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous immunoglobulins (IvIg) (Active Comparator): 3 x 0.36-0.44g/Kg IvIg every 4 weeks, then 3 months washing out, then 3x NaCl 0.9% every 4 weeks
  Interventions: Biological: intravenous immunoglobulins
- NaCl 0.9% (Placebo Comparator): NaCl 0.9%, 3x, every 4 weeks, then 3 months washing out, then 0.36-0.44g/Kg IvIg, 3x, every 4 weeks
  Interventions: Biological: intravenous immunoglobulins

INTERVENTIONS:
Biological: intravenous immunoglobulins — 0.36-0.44g/Kg IvIg intravenous, 3x, every 4 weeks
  Other Names: Gamunex 10%

SUMMARY:
The purpose of this study is to determine whether intravenous immunoglobulins are effective in the treatment of complex-regional pain syndrome.

DETAILED DESCRIPTION:
CRPS, a chronic pain syndrome associated with trophic disturbances is a frequent complication after limb trauma. More than one third of the CRPS will continue to chronic disease including loss of function in one limb. Some reports implicate an autoimmune pathogenesis of CRPS. Especially the finding of autoantibodies against peripheral neurons and successful treatment in single cases provide evidence for a possible successful treatment of CRPS with intravenous immunoglobulins (IvIg). Therefore IvIg may be an important anti-inflammatory treatment to prevent severe chronification of CRPS. Since IvIg is mainly effective in B-cell-mediated autoimmune diseases, autoantibodies against autonomic neurons and the concentration of B-cell activating factors BAFF and APRIL will be measured in the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* CRPS 1 (according to the IASP criteria) between 6 weeks and 6 months after diagnosis
* skin temperature of the affected side equal or higher than on non-affected side
* no change of the analgetic or co-analgetic medication within the last 10 days

Exclusion Criteria:

* Immunosuppressive or immunomodulatory treatment within the last three months
* CRPS previously treated with sympathetic block, lidocaine patch, local DMSO, spinal cord stimulation, intrathecal drug administration
* Known immune-mediated neuropathy (CIDP, MMN, MADSAM)
* Selective IgA-deficiency
* Severe heart disease
* Tumour disease in the last 5 years
* Allergy against Gamunex 10%
* Chronic renal disease Vaccination with live vaccine within the last three months
* Member of another clinical trial within the last 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-02-15 (Actual)

PRIMARY OUTCOMES:
Change in impairment Level SumScore (ISS) | after 0,3,6,9 months

SECONDARY OUTCOMES:
Pain disability score | 0,3,6,9 months
Quality of life (SF-36) | 0,3,6,9 months
Titer of surface-binding neuronal autoantibodies in the serum | 0,3,6,9 months
Serum concentration of B-cell activating factors BAFF, APRIL | 0,3,6,9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the Justus-Liebig-University, Giessen, Hesse, Germany

REFERENCES:
- [Background] Kohr D, Tschernatsch M, Schmitz K, Singh P, Kaps M, Schafer KH, Diener M, Mathies J, Matz O, Kummer W, Maihofner C, Fritz T, Birklein F, Blaes F. Autoantibodies in complex regional pain syndrome bind to a differentiation-dependent neuronal surface autoantigen. Pain. 2009 Jun;143(3):246-251. doi: 10.1016/j.pain.2009.03.009. Epub 2009 Apr 16. PMID 19375222
- [Background] Goebel A, Stock M, Deacon R, Sprotte G, Vincent A. Intravenous immunoglobulin response and evidence for pathogenic antibodies in a case of complex regional pain syndrome 1. Ann Neurol. 2005 Mar;57(3):463-4. doi: 10.1002/ana.20400. No abstract available. PMID 15732112